CLINICAL TRIAL: NCT01005979
Title: A Phase I Trial Using Cyclophosphamide, Rituximab and Revlimid (CR2) for the Treatment of Relapsed/Refractory B-Cell Chronic Lymphocytic Leukemia (B-CLL) and SLL
Brief Title: A Phase I Trial Using Cyclophosphamide, Rituximab and Revlimid (CR2) for the Treatment of Relapsed/Refractory B-Cell Chronic Lymphocytic Leukemia (B-CLL) and Small Lymphocytic Lymphoma (SLL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Emory University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Christopher R. Flowers, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00024085; WCI1642-09 (Other: Other)
Record Dates: First submitted 2009-09-30; First posted 2009-11-02 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Chronic Lymphocytic Leukemia; Lymphoma, Small Lymphocytic
Keywords: Leukemia, Lymphocytic, Chronic, B-Cell; Chronic Lymphocytic Leukemia; Lymphoma, Small Lymphocytic; Lymphoma; Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Leukemia | interventions — Lenalidomide; Rituximab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Lenalidomide, Rituximab, and Cyclophosphamide

INTERVENTIONS:
Drug: Lenalidomide, Rituximab, and Cyclophosphamide — COHORT 1: Cyclophosphamide 250 mg/m2 day 1, 2 and 3, Rituximab 500 mg/m2 i.v. day 1, Lenalidomide 2.5 mg/day starting day 8-28 of Cycle 1 and then daily on Days 1-28 of subsequent cycles
  COHORT 2: Cyclophosphamide 250mg/m2 day 1, 2 and 3. Rituximab 500 mg.m2 i.v. daY Lenalidomide 5 mg/day starting day 8 -28 of Cycle 1 and then daily on Days 1-28 of subsequent cycles
  COHORT 3: Cyclophosphamide 250mg/m2 day 1, 2 and 3, Rituximab 500 mg.m2 i.v. day 1, Lenalidomide 10 mg/day starting day 8 -28 of Cycle 1 and then daily on Days 1-28 of subsequent cycles
  COHORT 4: Cyclophosphamide 250mg/m2 day 1, 2 and 3, Rituximab 500 mg.m2 i.v. day 1, Lenalidomide 15 mg/day starting day 8 -28 of Cycle 1 and then daily on Days 1-28 of subsequent cycles
  Patients will receive a total of 6-8 cycles.
  Other Names: Revlimid; Rituxan; Mab Thera; Endoxan; Cytoxan; Neosar; Procytox; Revimmune

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD), safety and toxicity when cyclophosphamide, rituximab and lenalidomide (Revlimid) are combined for the treatment of relapsed/refractory of chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL).

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age ≥ 18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Relapsed/refractory B-cell CLL or SLL
5. All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 2 weeks prior to treatment in this study.
6. Patients must have received at least one prior therapy and must meet the NCI Working Group (NCI WG) Criteria for treatment of B-CLL as described in Appendix D.
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 at study entry (see Appendix C).
8. Laboratory test results within these ranges (unless related to CLL involvement):

   * Absolute neutrophil count ≥ 1000 /mm3
   * Platelet count ≥ 50,000/mm³
   * Serum creatinine ≤ 1.5 mg/dL. Serum creatinine > 1.5 mg/dL requires creatinine clearance of ≥ 60 mL/min by Cockroft-Gault formula.
   * Total bilirubin ≤ 1.5 mg/dL
   * Aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) ≤ 2 x upper limit of normal (ULN) or ≤ 5 x ULN if hepatic metastases are present.
9. Disease free of second malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.
10. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-International Units (mIU)/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix A: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods, AND also Appendix B: Education and Counseling Guidance Document.
11. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA] may use warfarin or low molecular weight heparin).

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Evidence of laboratory tumor lysis syndrome (TLS) by Cairo-Bishop criteria (Appendix J) (subjects may be enrolled upon correction of electrolyte abnormalities).
5. Use of any other experimental drug or therapy within 28 days of baseline.
6. Known hypersensitivity to thalidomide.
7. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
8. Any prior use of lenalidomide.
9. Concurrent use of other anti-cancer agents or treatments.
10. Known positive for HIV or infectious hepatitis, type A, B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to determine the maximum tolerated dose of lenalidomide in combination with cyclophosphamide and rituximab for the treatment of CLL or SLL. | Day 28 of the first cycle of chemotherapy

SECONDARY OUTCOMES:
Assess response criteria, including complete response rate, survival at 1 year, time to progression, duration of response, and eradication of minimal residual disease. | Response will be measured after 4 cycles, at the end of treatment and then every 3 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rajni Sinha, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States